CLINICAL TRIAL: NCT05926310
Title: Two-phase Pilot Study on the Safety and Feasibility of TWIICE Rise for Exoskeleton-assisted Ambulation in Patients With Spinal Cord Injury
Brief Title: Safety and Feasibility of TWIICE Rise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TWIICE (Industry)
Collaborators: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TWIICE_2021_15
Record Dates: First submitted 2023-06-06; First posted 2023-07-03 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-06

CONDITIONS: Spinal Cord Injuries; Gait Disorders, Neurologic
Keywords: Spinal Cord Injury; Exoskeleton; Robotics; Gait Rehabilitation; Lower-limb; Neurorehabilitation; Paraplegia; Walking; Assistive technology; Usability; Feasibility; Home use; Community use
MeSH Terms: conditions — Spinal Cord Injuries; Gait Disorders, Neurologic; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exoskeleton assisted ambulation (Experimental): Phase 1: Five participants will undergo a training programme with the TWIICE Rise 0.0 two times a week for up to 6 weeks for a total of 6 sessions.
  Phase 2: Ten participants will undergo a training programme with the TWIICE Rise 1.0 two times a week for up to 20 weeks for a total of 24 sessions.
  Interventions: Device: TWIICE Rise

INTERVENTIONS:
Device: TWIICE Rise — TWIICE Rise is a lower-limb overground robotic exoskeleton intended for patients with spinal cord injury (SCI).
  TWIICE Rise is intended to perform ambulatory functions in rehabilitation institutions, home, or community environment under the supervision of a specially trained coach.

SUMMARY:
The aim of this study is to assess the safety and the feasibility of two versions of TWIICE Rise for exoskeleton-assisted ambulation in patients with a spinal cord injury.

This study is done in two phases:

The first phase evaluates the safety and feasibility of TWIICE Rise 0.0 with 5 patients over 6 sessions in clinic. The second phase is being conducted with TWIICE Rise 1.0. This version has potentially improved functionalities based on feedback from Phase 1. Safety and feasibility will be assessed with 10 patients over 24 sessions in different settings (clinic, home, and community environment).

DETAILED DESCRIPTION:
The aim of this clinical trial is to assess the safety and the feasibility of two versions of TWIICE Rise for exoskeleton assisted ambulation in patients with a spinal cord injury. The study is thus done in two phases.

The first phase evaluates the safety and feasibility of TWIICE Rise 0.0 with five patients over 6 sessions in clinic. This phase allows the manufacturer to collect data that can be used to improve the device design if necessary.

The second phase of the study is being conducted with TWIICE Rise 1.0. Safety and feasibility will be assessed with 10 patients over 24 sessions in different settings (clinic, home, and community environment) to test the device intended use. The first sessions are done at the rehabilitation specialized center to benefit from the clinical settings to learn to walk with the exoskeleton. Once the patients reach sufficient ambulatory skills determined by a score of 29 in the Mobility SkillsTests, the following sessions can be done at home and community settings.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent signed by the subject.
2. Traumatic and non-traumatic SCI
3. Motor incomplete SCI with Neurological Level of Injury (NLI) C5-L5, or Motor Complete SCI with NLI T1-L5 as determined by the ISNCSCI.
4. Male and non-pregnant, non-lactating female aged 18 to 70 years old
5. At least 6 months after injury
6. Able to stand or maintain upright position with a standing device (e.g., 'Easy stand') for at least ten minutes without clinical symptoms of orthostatic hypotension.
7. Able to use crutches.
8. Able to sit with knees and hips >= 90° flexion
9. Phase 1: Height of 160 to 180 cm, Phase 2: Height of 160 to 190 cm
10. Phase 1: Weight of <80 kg, Phase 2: Weight of <100 kg

Exclusion Criteria:

1. History of severe neurological injuries other than spinal cord injury (e.g., Multiple Sclerosis, Cerebral Palsy, Amyotrophic Lateral Sclerosis, Traumatic Brain Injury, Stroke)
2. Ability to walk 10 meters without physical assistance of a person
3. Severe concurrent medical disease, illness, or condition
4. Systemic or peripheral infection influencing wearing an exoskeleton.
5. Diagnosis of coronary artery disease that precludes moderate to intense exercise.
6. A medical diagnosis in the patient chart of atherosclerosis, congestive heart failure, or history of myocardial infarction
7. Individuals with a pacemaker, defibrillator, drug delivery pump, or other electrical devices if malfunctions could lead to serious adverse events.
8. Deep vein thromboses in lower extremities of less than 6 months duration.
9. Untreated sever hypertension (systolic blood pressure >180 mmHg, diastolic blood pressure >120 mmHg)
10. Unstable spine or unhealed limbs
11. History of lower extremities or pelvic fragility fractures within the last two years
12. Heterotopic ossification that impairs joint mobility
13. Significant contractures defined as flexion contracture limited to 20 the hip and knee.
14. Severe spasticity (Modified Ashworth grade 4) or uncontrolled clonus
15. Diagnosis of severe osteoporosis/penia: Dual Energy X-ray Absorptiometry (DXA) results indicating a t-score below -3.5 at the femoral neck or the total proximal femur bone, and knee bone mineral density (BMD) < 0.60 gm/cm2
16. Current pressure ulcer of the arms, trunk, pelvic area, or lower extremities
17. Psychiatric or cognitive conditions that may interfere with the trial.
18. Pregnancy or women who plan to become pregnant during the study period, and lactating women.
19. Patient is currently involved in any other interventional study.
20. Other severe illness that the study physician considers in his/her clinical judgment to be exclusionary.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of (serious) adverse device effects [Safety] | up to 26 weeks
  This outcome is commonly used in healthcare for the measurement of patient safety.
Incidence of device deficiency [Safety] | up to 26 weeks
  This outcome is commonly used in healthcare for the measurement of patient safety.

SECONDARY OUTCOMES:
Incidence of (serious) adverse events [Safety] | up to 26 weeks
  This outcome is commonly used in healthcare for the measurement of patient safety.
Heart rate (pre-training, when standing, and post-training) [Safety] | up to 10 weeks
  Used to assess whether significant changes in essential physiological functions occur following training with TWIICE Rise.
Systolic and diastolic blood pressure (pre-training, when standing, and post-training) [Safety] | up to 10 weeks
  Used to assess whether significant changes in essential physiological functions occur following training with TWIICE Rise.
Pain rating and location [Safety] | up to 26 weeks
  Used to assess whether training with TWIICE Rise does not cause or exacerbate pain.
  Pain intensity and location are assessed at the beginning of each session. Pain intensity is evaluated using the Pain Numeric Rating Scale that is a unidimensional measure of pain in adult. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Fatigue rating [Safety] | up to 26 weeks
  Used as a measure of exertion due to training with TWIICE Rise. Fatigue is assessed pre-training and post training. The Fatigue Numeric Rating Scale is a patient-administered, single-item, 11-point horizontal scale anchored at 0 and 10, with 0 representing 'no fatigue' and 10 representing 'as bad as you can imagine'.
Skin status rating [Safety] | up to 26 weeks
  Used to assess whether the device's interfaces cause skin lesions. Skin status is rated on a 0 to 4 pressure ulcer scale, 0 representing 'no skin injury' and '4' representing 'very deep wound'.
Number of steps taken [Feasibility] | up to 26 weeks
  TWIICE Rise will record the number of steps, walking time, standing time, and walking distance, step frequency, mid-stride pause every session. This information will allow insight into the proportion of time spent training per session.
Training location [Feasibility, phase 2 only] | up to 26 weeks
  Used to evaluate the feasibility of using the device in different environments such clinics, home and community settings and the number of sessions in each condition
Type of suface walked on [Feasibility] | up to 26 weeks
  This indicated the feasibility of walking on different type of terrain.
6-Meter Walk Test (6MWT) + Level of Assistance [Feasibility] | up to 26 weeks
  The distance walked with the powered exoskeleton during the 6MWT. The 6MWT is the primary assessment used to determine the progression of walking skills in exoskeletons.
10-Meter Walk Test (10MWT) + Level of Assistance [Feasibility] | up to 26 weeks
  The 10MWT is the best effort time (seconds) it takes the participant to walk a 10 m distance and is recorded while the person performs the 6MWT. This allows assessing the walking speed.
Time Up and Go (TUG) + Level of Assistance [Feasibility] | up to 26 weeks
  The TUG test measures the time it takes the participant to stand up from a seated position, walk three meters, turn around, walk back, and sit down again. The TUG test represents the person s ability to use the exoskeletal system since it incorporates multiple aspects of mobility in the device.
Donning and doffing time + Level of Assistance [Feasibility] | up to 26 weeks
  Used to evaluate the time needed to install the user inside the device (donning) and back to the wheelchair (doffing). It assesses the feasibility and usability of a device, as the setup time is usually a determining factor for assisting devices.
Mobility skills test + Level of Assistance [Feasibility] | up to 26 weeks
  Used to assess the feasibility of the mobility tasks intended with TWIICE Rise. Mobility skills such as standing, walking on different type of ground, and step on a stair are measured separately of each other in an ascending order of difficulty, until two skills cannot be achieved without moderate or maximal assistance.

OTHER OUTCOMES:
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) [Satisfaction] | up to 26 weeks
  Used to measure user satisfaction from participants and therapists. The Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) is designed to measure the level of satisfaction and the value people attribute to assistive technologies. It does so using 12 variables which are scored on a 5 point scale in terms of perceived importance and satisfaction. While items 1-8 rate the satisfaction with the device, items 9-12 are for assessing the satisfaction with the service. If the users are not very satisfied with a feature, they are asked to provide specific feedback. The final score is the mean sum scores of all valid responses with a range of 1 (not satisfied at all) to 5 (very satisfied).
Open-ended questionnaire [Satisfaction] | up to 26 weeks
  Used to study design modifications requested by users and clinicians.
Subjective health-related questionnaire [General Health] | up to 26 weeks
  4-item questionnaire to assess potential health-related changes due to regular exoskeleton-assisted ambulation, with a 5-point Likert-scale (1 = 'strongly disagree' and 5 = 'strongly agree').
Psychosocial Impact of Assistive Devices Scales [General Health] | up to 26 weeks
  The Psychosocial Impact of Assistive Devices Scales (PIADS) is a 26-item (7-point Likert-Scale), self-report questionnaire designed to assess the effects of an assistive device on functional independence, well-being, and quality of life. It is divided into three subscales: Competence, adaptability and self-esteem. For each of the subscales, typically means are calculated that range from -3 (maximum negative impact) to +3 (maximum positive impact). To have only positive sum scores, the range of the individual scores are shifted to 1 to 7, meaning that sum scores range from 1 *26 (26, maximum negative impact) to 7 *26 (182, maximum positive impact). The PIADS is a responsive measure and sensitive to important variables such as the user's clinical condition, device stigma, and functional features of the device. It has been shown to accurately reflect the self-described experiences of people who use assistive devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre Nottwil, Nottwil, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Lang C, Eriks-Hoogland I, Perret C, Bouri M, Widmer M. Safety assessment and feasibility of the TWIICE powered exoskeleton for assisted ambulation in individuals with spinal cord injury. J Neuroeng Rehabil. 2025 Sep 26;22(1):194. doi: 10.1186/s12984-025-01727-4. PMID 41013571